CLINICAL TRIAL: NCT03408873
Title: Enhancing Adherence and Outcomes in Bipolar Disorder With Abilify Maintena + a Targeted Behavioral Approach to Promote Sustained Adherence and Behavioral Change
Brief Title: CAE Plus LAI in Individuals With Bipolar Disorder at Risk for Treatment Non-adherence (BD-CAEL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Martha Sajatovic (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I0113
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Bipolar Disorder; Medication Adherence; Medication Non Adherence
Keywords: Antipsychotic Drugs; Antipsychotics; Injectables; Long Acting Injectable Antipsychotic; Bipolar Disorder; Medication Adherence; Medication Non-Adherence
MeSH Terms: conditions — Bipolar Disorder; Medication Adherence | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Noncompliance (Experimental): Subjects enrolled in the study will receive both Abilify Miantena and the Customized Adherence Enhancement (CAE) intervention
  Interventions: Drug: Abilify Maintena; Behavioral: Customized Adherence Enhancement (CAE)

INTERVENTIONS:
Drug: Abilify Maintena — Drug is in an injectable form and will be administered approximately every four weeks through Week 24 of the study. Dosage is per package insert or at the discretion of the psychiatrist.
Behavioral: Customized Adherence Enhancement (CAE) — CAE targets key areas relevant to non-adherent populations with schizophrenia or schizoaffective disorder: 1) inadequate or incorrect understanding of mental disorder; 2) lack of medication-taking routines; 3) poor communication with care providers; and 4) substance use which interferes with adherence and healthy behaviors that promote recovery. CAE is delivered based upon initial assessment of reasons for non-adherence and only those components of CAE that are determined to be indicated for that individual are delivered (psychoeducation, modified motivational interviewing, assistance with medication routines, coaching in communication with providers).

SUMMARY:
This is a prospective study using customized adherence enhancement (CAE) and long-acting injectable (LAI) antipsychotic in 30 individuals with bipolar disorder (BD) at risk for treatment non-adherence. The CAE approach is expected to improve treatment adherence, as well as improve BD symptoms, functioning and treatment attitudes among subjects with bipolar disorder.

DETAILED DESCRIPTION:
Oral Abilify (aripiprazole) is effective in the treatment of patients with BD when prescribed as an acute anti-manic agent and for the maintenance treatment of bipolar disorder. Abilify Maintena is an intramuscular (IM) depot formulation of oral aripiprazole (Abilify). Abilify Maintena appears to be as effective as standard oral Abilify and may maximize patient adherence. Recent clinical trials suggest that Abilify Maintena is effective for the treatment of patients with BD.

Customized Adherence Enhancement (CAE) is a brief behavioral intervention that improves adherence approximately 30% more than an educational control in adults with BD. The CAE program is a brief, practical intervention consisting of a series of up to four psychosocial treatment modules based upon an adult's unique adherence barriers: 1) Psychoeducation on BD Medications; 2) Communication with Providers; 3) Strategies to Enhance Medication Routines; and 4) Targeting Substance Use Problems with Modified Motivational Enhancement Therapy. Multiple studies conducted by these investigators has shown that CAE is effective in in treating poorly adherent BD adults.

In addition, studies by these investigators have shown that combining LAI + CAE dramatically improves adherence, symptoms and functional outcomes in people with schizophrenia and schizoaffective disorder. In summary, LAI can maximize medication adherence, while CAE addresses individual barriers to sustained adherence and behavioral change. Combining LAI + CAE improves adherence, symptoms and functioning in high-risk people with primary psychotic disorders. The proposed project will test the efficacy of combining Abilify Maintena with CAE to help improve outcomes in poorly adherent patients with BD. Pilot data suggest that adherence with concomitantly prescribed psychotropic drugs improves with LAI + CAE. The findings have particular relevance to BD because many BD patients are on concomitant oral psychotropic drugs in addition to antipsychotic. Thus, it is expected that combining CAE with LAI will lead to a "halo effect" in that these BD patients will engage in their own care more broadly.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals age 18 and older with BD Type 1 or 2 as confirmed by the Mini International Psychiatric Inventory (MINI).
2. Known to have medication treatment adherence problems as identified by the Treatment Routines Questionnaire (TRQ, 20% or more missed medications in past week or past month)
3. Screening the Brief Psychiatric Rating Scale (BPRS) score of ≥ 36
4. Ability to be rated on psychiatric rating scales.
5. Willingness to take long-acting injectable antipsychotic medication (LAI)
6. Currently in treatment or scheduled to receive treatment at a Community Mental Health Clinic (CMHC) or other clinical setting able to provide mental health care during and after study participation
7. Able to provide written, informed consent to study participation.

Exclusion Criteria:

1. Individuals on LAI immediately prior to study enrollment.
2. Individuals with known intolerance or resistance to either oral aripiprazole or LAI formulation of aripiprazole
3. Prior or current treatment with clozapine
4. Medical condition or illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial
5. Physical dependence on substances (alcohol or illicit drugs) likely to lead to withdrawal reaction during the course of the study in the clinical opinion of the treated research psychiatrist
6. Immediate risk of harm to self or others
7. Female who is currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Sajatovic M, Levin JB, Ramirez LF, Cassidy KA, McNamara N, Fuentes-Casiano E, Wilson B, Appling D, S FB. Long-Acting Injectable Antipsychotic Medication Plus Customized Adherence Enhancement in Poor Adherence Patients With Bipolar Disorder. Prim Care Companion CNS Disord. 2021 Sep 16;23(5):20m02888. doi: 10.4088/PCC.20m02888. PMID 34534421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: . Individuals were recruited from an academic medical center and via outreach to community settings including community mental health clinics (CMHCs). Enrolled participants had self-reported adherence problems as identified by the TRQ (≥20% missed BD medications in past week or past month), a screening Brief Psychiatric Rating Scale15 score ≥36, willingness to take LAI, and were in treatment at a CMHC or other clinical setting.
  Participants were adults ≥ age 18 with Type 1 or Type 2 BD.
Groups:
- CAE-L: Subjects enrolled in the study will receive both Abilify Miantena and the Customized Adherence Enhancement (CAE) intervention
  Abilify Maintena: Drug is in an injectable form and will be administered approximately every four weeks through Week 24 of the study. Dosage is per package insert or at the discretion of the psychiatrist.
  Customized Adherence Enhancement (CAE): CAE targets key areas relevant to non-adherent populations with schizophrenia or schizoaffective disorder: 1) inadequate or incorrect understanding of mental disorder; 2) lack of medication-taking routines; 3) poor communication with care providers; and 4) substance use which interferes with adherence and healthy behaviors that promote recovery. CAE is delivered based upon initial assessment of reasons for non-adherence and only those components of CAE that are determined to be indicated for that individual are delivered (psychoeducation, modified motivational interviewing, assistance with medication routines, coaching in communication with providers).
Period: Visit 1 Assessment (Baseline)
Arm/Group | CAE-L
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3
Period: Visit 2 Assessment
Arm/Group | CAE-L
Started | 27
Completed | 26
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Visit 3 Assessment
Arm/Group | CAE-L
Started | 26
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Visit 4 Assessment
Arm/Group | CAE-L
Started | 25
Completed | 23
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Visit 5 Assessment
Arm/Group | CAE-L
Started | 23
Completed | 22
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Visit 6 Assessment
Arm/Group | CAE-L
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Visit 7 Assessment
Arm/Group | CAE-L
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CAE-L
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.47 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Black or African American | 17
  Other or Multiracial | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1
  Non Hispanic | 29
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 17
  Married | 1
  Separated/Divorced/Widowed | 12
Mean Years of Education Attained [Mean (Standard Deviation); unit: years] | 13.63 (2.85)
Occupation Status [Count of Participants; unit: Participants]
  Full time employment/homemaker | 0
  Part time employment/ homemaker or student | 4
  Unemployed or on disability | 25
  Other | 1
Number of Participants Who Live Alone [Count of Participants; unit: Participants] | 16
Age at Bipolar onset [Mean (Standard Deviation); unit: years] | 27.63 (11.80)
Duration of bipolar illness [Mean (Standard Deviation); unit: years] | 21.56 (11.74)
Number of Participants With Current Substance Use Problems [Count of Participants; unit: Participants] — Non-alcohol Substance Use Disorder from the past 12 months derived from the Mini-International Neuropsychiatric Interview (MINI) diagnostic interview for the major psychiatric disorders in DSM-III-R, DSM-IV and DSM-5 and ICD-10.
  Participants | 6
Mean lifetime psychiatric hospitalizations [Mean (Standard Deviation); unit: hospitalizations] | 3.07 (3.43)
Mean lifetime substance abuse hospitalizations [Mean (Standard Deviation); unit: hospitalizations] | 1.06 (2.00)
Number of Participants With History of Physical Abuse [Count of Participants; unit: Participants] | 16
Number of Participants With History of Sexual Abuse [Count of Participants; unit: Participants] | 10
Number of Participants With Family history of Mental Illness [Count of Participants; unit: Participants] | 28
Number of Participants With Family history of Substance Abuse [Count of Participants; unit: Participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Tablets Routine Questionnaire (TRQ, Past Week)
Description: Treatment non-adherence is measured as a percentage of medications not taken within the past week at time of assessment.
  The minimum score is 0% and the maximum score is 100%. A higher score implies poorer treatment adherence.
Time Frame: Screen to Week 24
Population: Poorly adherent patients with bipolar disorder who received long-acting injectable antipsychotic medication and a customized adherence enhancement intervention (CAE).
  Descriptive statistics (means and standard deviations or counts and percentages) were generated for all outcomes measures using complete cases.
Measure: Mean (Standard Deviation); unit: percentage of missed BD medications
Arm/Group | CAE-L
Number analyzed (Participants) | 29
percentage of missed BD medications
  Screen | 50.1 (24.8)
  Baseline: number analyzed (Participants) | 28
  Baseline | 37.5 (30.0)
  Week 24: number analyzed (Participants) | 11
  Week 24 | 16.9 (26.97)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between screen & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 29 participants with screen data only 11 had Week 24 data. Statistical Analysis was conducted for 11 participants with data at the 2 timepoints. Thus, the mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -31.4
Statistical Analysis 2: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between baseline & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 28 participants with baseline data only 11 had Week 24 data. Statistical Analysis was conducted for 11 participants with data at the 2 timepoints. The mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p = 0.12, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -11.7

2. Primary Outcome: Change in Tablets Routine Questionnaire (TRQ, Past Month)
Description: Treatment non-adherence is measured as a percentage of medications not taken within the past month at time of assessment.
  The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of missed BD medications
Arm/Group | CAE-L
Number analyzed (Participants) | 29
percentage of missed BD medications
  Screen | 40.6 (23.7)
  Baseline: number analyzed (Participants) | 28
  Baseline | 29.4 (21.6)
  Week 24: number analyzed (Participants) | 11
  Week 24 | 19.2 (24.5)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0599, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -19.6
Statistical Analysis 2: Comparison: CAE-L; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.63, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.2

3. Primary Outcome: LAI Injection Adherence
Description: LAI injection adherence will be determined as a proportion of LAI injections received at the appropriate time (within 7 days of scheduled time).
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | CAE-L
Number analyzed (Participants) | 20
percentage of adherence | 100 (0)

4. Secondary Outcome: Change in the Brief Psychiatric Rating Scale (BPRS) Score
Description: The BPRS measure psychiatric symptoms such as depression, anxiety, hallucinations and unusual behavior. The minimum score is 18 and the maximum score is 126. A higher score implies a worse condition.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Baseline | 36.4 (7.4)
  Week 24: number analyzed (Participants) | 19
  Week 24 | 24.9 (5.7)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between baseline & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 30 participants with baseline data only 19 had Week 24 data. Statistical Analysis was conducted for 19 participants with data at the 2 timepoints. The mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -10.7

5. Secondary Outcome: Change in Young Mania Rating Scale (YMRS) Score
Description: The YMRS measures symptoms of mania. The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 13.2 (6.2)
  Baseline | 10.4 (5.6)
  Week 24: number analyzed (Participants) | 19
  Week 24 | 5.6 (4.3)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between screen & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 30 participants with screen data, only 19 had Week 24 data. Statistical Analysis was conducted for 19 participants with data at the 2 timepoints. Thus, the mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -8.4
Statistical Analysis 2: Comparison: CAE-L; We compared for the primary and secondary outcomes across two sets of time-points: 1) difference between screen and week 24, and 2) between baseline and week 24. A non-parametric Wilcoxon signed-rank test compared these repeated measurements (matched on participant) between these time-points to determine whether the population medians differed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -5.8

6. Secondary Outcome: Change in Montgomery Asberg Rating Scale (MADRS) Score
Description: The MADRS measures symptoms of depression. The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 24.5 (5.7)
  Baseline | 18.1 (9.4)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 7.95 (8.2)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between screen & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 30 participants with screen data, only 21 had Week 24 data. Statistical Analysis was conducted for 21 participants with data at the 2 timepoints. Thus, the mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -16.6
Statistical Analysis 2: Comparison: CAE-L; [analysis description as in outcome 5, analysis 2]; Test type: Other — We compared the repeated measure outcome across 2 time-points (difference between baseline & week 24) to determine whether the population medians differed matched on participant with complete data. Of the 30 participants with baseline data, only 21 had Week 24 data. Statistical Analysis was conducted for 21 participants with data at the 2 timepoints. The mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; p = 0.003, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -8.1

7. Secondary Outcome: Change in Clinical Global Impressions (CGI) Score
Description: The minimum possible score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen: number analyzed (Participants) | 29
  Screen | 4.6 (0.5)
  Baseline | 4.1 (0.6)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 2.8 (0.8)
Statistical Analysis 1: Comparison: CAE-L; Test type: Other — We compared the repeated measure outcome across 2 time-points (difference between screen & week 24 to determine whether the population medians differed matched on participant with complete data; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.8
Statistical Analysis 2: Comparison: CAE-L; We compared for the primary and secondary outcomes across two time-points: difference between baseline and week 24. A non-parametric Wilcoxon signed-rank test compared these repeated measurements (matched on participant with complete data) between these time-points to determine whether the population medians differed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.3

8. Secondary Outcome: Change in Drug Attitude Inventory (DAI) Score
Description: DAI-10 scoring ranges from -10 to +10 with a total score >0 indicating a positive attitude toward psychiatric medications and a total score of <0 indicating a negative attitude toward psychiatric medications
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 7.2 (1.9)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 8.1 (1.4)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 5, analysis 2]; Test type: Other; p = 0.0566, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.8

9. Secondary Outcome: Change in Attitude Towards Medication Questionnaire (AMSQ) Score
Description: A modification of the Lithium Attitudes Questionnaire (Harvey 1991) which evaluates an individual's attitudes towards mood stabilizers. The AMSQ is used to measure attitudes towards medications. The scale contains 19 items grouped into 7 subscales: general opposition to prophylaxis (4 items), denial of therapeutic effectiveness (2 items), fear of side effects (2 items), difficulty with medication routines (4 items), denial of illness severity (3 items), negative attitudes toward drugs in general (3 items), and lack of information about psychiatric medication (1 item). Responses which suggest positive attitudes towards medications are scored "0", while responses which suggest negative attitudes towards medications are scored "1". The items scores are added for a total score which is reported, with the minimum total score of 0 and maximum total score of 19. Higher scores on each subscale represent more negative attitudes toward mood stabilizers.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 7.9 (3.3)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 4.0 (3.4)
Statistical Analysis 1: Comparison: CAE-L; We compared for the primary and secondary outcomes across two time-points: difference between screen and week 24. A non-parametric Wilcoxon signed-rank test compared these repeated measurements (matched on participant with complete data) between these time-points to determine whether the population medians differed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.4

10. Secondary Outcome: Change in Social and Occupational Functioning Assessment Scale (SOFAS) Score
Description: The SOFAS measures social and occupational functioning independent of the overall severity of the individual's psychological symptoms. The minimum score is 0 and the maximum score is 100. A higher rating implies a higher level of functioning.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Baseline | 51.9 (8.1)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 70.8 (8.1)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 6, analysis 1]; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 17.7

11. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Score
Description: The minimum score is 1 and the maximum score is 100. A higher score implies higher functioning.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Baseline | 53.5 (8.1)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 70.7 (7.9)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between baseline & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 30 participants with baseline data, only 21 had Week 24 data. Statistical Analysis was conducted for 21 participants with data at the 2 timepoints. The mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 16.9

12. Secondary Outcome: Change in Oxford Bipolar Knowledge Questionnaires (OBQ) Score
Description: The OBQ assess knowledge of BD management. Total score rangers from 0-80, with a higher score indicative of better knowledge of bipolar mood management.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 29
score on a scale
  Screen | 52.9 (16.1)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 70.7 (8.4)
Statistical Analysis 1: Comparison: CAE-L; We compared the repeated measure outcome across 2 time-points (difference between screen & week 24 to determine whether the population medians differed matched on participant with complete data. Of the 29 participants with screen data, only 21 had Week 24 data. Statistical Analysis was conducted for 21 participants with data at the 2 timepoints. Thus, the mean difference reported is not consistent with the mean values reported because only those with complete data were included in the analysis; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 14.7

13. Secondary Outcome: Change in The Self-Report Habit Index (SRHI) Score
Description: The SRHI is a measure of habit strength. The minimum score is 12 and the maximum score is 84. A higher score implies stronger habits.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 47.3 (12.4)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 68.5 (13.8)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 6, analysis 1]; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 19.2

14. Secondary Outcome: Change in Communication Styles Scale Score
Description: The Communication Styles Scale is a measure of the impact of physician communication style on medication beliefs and adherence behavior. Total scores range from 0-27 where the higher score indicates a more initial collaborative communication style.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 22.4 (4.2)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 22.1 (6.3)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.73, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.5

15. Secondary Outcome: Change in Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES 8A) Score
Description: The SOCRATES measures motivation to reduce the use of substances. The minimum score is 10 and the maximum score is 50. A higher score indicates a higher desire to reduce drinking.
Time Frame: Screen to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAE-L
Number analyzed (Participants) | 30
score on a scale
  Screen | 46.8 (16.8)
  Week 24: number analyzed (Participants) | 21
  Week 24 | 34.8 (18.7)
Statistical Analysis 1: Comparison: CAE-L; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -10.7

ADVERSE EVENTS:
Time Frame: Safety evaluations at baseline & Week 24 included basic laboratory evaluations (comprehensive metabolic panel, lipid profile, complete blood count (CBC) with differential & pregnancy testing).EKGs at baseline & Weeks 4 & 24. Side effects, vital signs & weight assessed at each clinical visit &standardized measures of extrapyramidal symptoms i.e.Simpson Angus Scale (SAS)Barnes Akathisia Scale(BAS) Abnormal Involuntary Movement Scale(AIMS) &Extrapyramidal Symptoms Scale-Abbreviated version(ESRS-A).
Arm/Group | CAE-L
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 23/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CAE-L (N=30)
Injection site pain or reaction (Skin and subcutaneous tissue disorders) | 7/23
Drowsiness (Nervous system disorders) | 7/23
Tremor (Nervous system disorders) | 6/23
Sexual dysfunction (Reproductive system and breast disorders) | 3/23
Drooling (General disorders) | 2/23
Muscle Movement complaints (Musculoskeletal and connective tissue disorders) | 2/23
Weight gain (Metabolism and nutrition disorders) | 2/23

LIMITATIONS AND CAVEATS:
This study had a number of limitations including small sample, non-controlled design, and single-site setting. An additional limitation is that adherence was based upon self-report, which has potential to under-count missed medication. The improvement in adherence behaviors immediately after screen (and before CAE was administered) may possibly reflect a Hawthorne effect which could have obscured improvement in CAE-related change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03408873/Prot_SAP_000.pdf